CLINICAL TRIAL: NCT04331847
Title: AMoCo Study: Abortion-related Morbidity and Mortality in Conflict-affected and Fragile Settings Study
Brief Title: Abortion-related Morbidity and Mortality in Conflict-affected and Fragile Settings Study
Acronym: AMoCo
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Epicentre (Other)
Collaborators: Ipas (Other); Guttmacher Institute (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: Elrha-R2HC; 509 (Other: Guttmatcher Institute); 18110 (Other: MSF ERB)
Record Dates: First submitted 2020-01-14; First posted 2020-04-02 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-06

CONDITIONS: Abortion Complication
Keywords: Near-miss; Risks factors; Maternal health; Abortion; Maternal mortality
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Quantitative observational descriptive study: among women presenting for abortion-related complications
- Qualitative study: among women with a near-miss or a potentially life-threatening complication
- Rapid health facility assessment with the health professional: in charge of Post-Abortion Care
- Knowledge Attitudes, Practice and Behavior quantitative survey: among health care providers involved in the management of abortion-related complications

SUMMARY:
To describe and estimate the burden of abortion-related complications, particularly near-miss complications and deaths, and their associated factors among women presenting for abortion-related complications in health facilities supported by Médecins Sans Frontières (MSF) in African fragile and/or conflict-affected settings.

DETAILED DESCRIPTION:
Multi-sites mixed-methods study with 4 components:

1. A quantitative observational descriptive study among women presenting for abortion-related complications to determine the frequency and severity of abortion-related complications including near-miss cases and death. Data will be collected through a medical records review and a quantitative survey among women presenting for abortion-related complications to determine the sociodemographic and clinical characteristics of the women with abortion-related complications, the type of abortion, the type and severity of complications and the clinical management received. It will also give insight into the characteristics of near-miss events following unsafe abortion.
2. A qualitative study about women's experiences associated with a near-miss event (and potentially life threatening): their pathway of access to care including their decision-making process, their own perceptions and opinions and other factors or conditions that might contribute to the near-miss event (in-depth face to face interviews).
3. A rapid health facility assessment with the health professional in charge of Post-Abortion Care will complement the assessment of the quality of management of complications
4. A Knowledge Attitudes, Practice and Behavior quantitative survey among health care providers involved in the management of abortion-related complications will identify provider-associated factors that may contribute to near-miss events.

ELIGIBILITY:
MEDICAL RECORD REVIEW:

Inclusion Criteria:

Women

* with any signs or symptoms of abortion-related complications, i.e. any signs or symptoms of complications of spontaneous or induced abortion, whatever the abortion stage: inevitable, missed, incomplete, complete abortion .
* Or with a presentation primary diagnosis of ectopic pregnancy or molar pregnancy

Exclusion Criteria:

* Threatened abortion (defined as vaginal bleeding with a closed cervix after having excluded the diagnosis of ectopic pregnancy or molar pregnancy)
* History of abortion-related complications and presenting for an unrelated issue
* Refusal to participate

QUANTITATIVE INTERVIEW:

Inclusion criteria: all women included in the medical record review subcomponent and hospitalized (who stayed overnight or more)

Exclusion criteria:

Participation to the interview as potentially harmwful to the woman according to her health care provider, Refusal to participate.

QUALITATIVE INTERVIEW:

Inclusion criteria: Women eligible for the quantitative interview and who experienced at least 1 criterion of near-miss event or potentially life-threatening conditions

Exclusion criteria:

Participation to the interview as potentially harmwful to the woman according to her health care provider, Refusal to participate.

RAPID FACILITY ASSESSMENT:

Key-informant: the provider in charge of the service providing post-abortion care

KAPB SURVEY:

Inclusion criteria:

Health professionals (i.e. doctors, midwives, clinical officers, medical officers, nurses, aidmidwives, aid-nurses) involved in PAC and SAC services in the study site health facility Literate

Exclusion criteria:

Refusal to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women presenting to the wards of the study sites which see women presenting for PAC (emergency unit, gyn/obs units, ICU unit, PAC unit, etc. according to site).
  The provider in charge of the service providing post-abortion care, in each study sites, will be the key-informant who will answer the rapid facility assessment questionnaire.
  All health professionals involved in PAC and SAC services will be proposed to participate in the KAPB survey
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
From the Quantitative observational descriptive study: | Between september 2019 and February 2021
  Proportion of near-miss cases among all women presenting for abortion-related complications.

SECONDARY OUTCOMES:
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Facility-based abortion-related complications ratio per annum for the following denominators: live births, all admissions and deliveries
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Facility-based abortion-related near-miss ratio per annum for the following denominators: live births, abortion-related admissions, all admissions and deliveries
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Facility-based abortion-related mortality ratio per annum for the following denominators: live births, abortion-related admissions, all admissions and deliveries
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Facility-based abortion-related severe maternal outcome ratio: the number of women with severe abortion-related maternal outcome (near-miss + death) per 1000 live births (LB)
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Facility-based abortion-related near-miss mortality ratio: ratio between abortion-related near- miss cases and abortion-related deaths
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Facility-based abortion-related mortality index : number of abortion-related maternal deaths divided by the number of women with abortion-related severe maternal outcome expressed as a percentage
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Proportional morbidity: proportion of each type of abortion-related complication among all complications
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Proportion of women disclosing or presenting signs of induced abortion attempt
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Proportion of each induced abortion method used
Quantitative observational descriptive study: medical record review+quantitative interviews: | Between september 2019 and February 2021
  Risk factors (socio-demographic characteristics, obstetrical history, induced abortion, displacement/exposure to conflict, exposure to violence, delay in accessing care) associated with abortion related near-miss events
Qualitative study (qualitative in-depth interviews): | Between september 2019 and February 2021
  Description of the woman pathway to care
Qualitative study (qualitative in-depth interviews): | Between september 2019 and February 2021
  Description of perceptions and opinions about their own experience
Qualitative study (qualitative in-depth interviews): | Between september 2019 and February 2021
  Description of conditions and factors that could contribute to the potentially life-threatening conditions and near-miss event.
Knowledge Attitude Practice and Behavior (KAPB) survey: | Between september 2019 and February 2021
  Proportion of each knowledge, attitude and practice of health facility staff related to Post Abortion Care and Safe Abortion Care

CONTACTS AND LOCATIONS:
Overall Officials: FETTERS Tamara, Study Director — Ipas; PASQUIER Estelle, Study Director — Epicentre
Locations (3):
- Castor Maternity Center, Bangui, Central African Republic
- Maternity center of the Hopital General de Référence, Masisi, Democratic Republic of the Congo
- Maternity center of the general Jahun Hospital, Jahun, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
A Memorandum of Understanding includes a chapter on data sharing agreement (DSA) between each of the partners (MSF-Epicentre/Ipas/Guttmacher) has been signed.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From June 2020 to December 2021
Access Criteria: Partners of the study